CLINICAL TRIAL: NCT02010606
Title: Phase I Trial of Vaccination With Autologous Dendritic Cells Pulsed With Lysate Derived From an Allogeneic Glioblastoma Stem-like Cell Line for Patients With Newly Diagnosed or Recurrent Glioblastoma
Brief Title: Phase I Study of a Dendritic Cell Vaccine for Patients With Either Newly Diagnosed or Recurrent Glioblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Jethro Hu, Faculty Neuro-Oncologist, Cedars-Sinai Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 33203
Record Dates: First submitted 2013-12-02; First posted 2013-12-13 (Estimated); Last update posted 2021-11-22 (Actual); Status verified 2021-11

CONDITIONS: Glioblastoma; Glioblastoma Multiforme; Glioma; Astrocytoma; Brain Tumor
Keywords: Newly diagnosed glioblastoma; Recurrent glioblastoma; Dendritic cell vaccine; Immunotherapy; Cancer stem cells; Glioma stem cells; Glioma stem-like cells; Cancer stem-like cells; Neurosphere; Therapeutic Uses; Antineoplastic Agents; Neoplasms; Immunologic Factors; Interferon Inducers; Physiological Effects of Drugs; Pharmacologic Actions
MeSH Terms: conditions — Glioblastoma; Glioma; Astrocytoma; Brain Neoplasms; Neoplasms | interventions — Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort A: Patients with newly diagnosed glioblastoma (Experimental): Dendritic cell vaccination, in addition to standard temozolomide chemotherapy and involved field radiation therapy
  Interventions: Biological: Dendritic cell vaccination, in addition to standard temozolomide chemotherapy and involved field radiation therapy
- Cohort B: Patients with recurrent glioblastoma (Experimental): Dendritic cell vaccination, with optional bevacizumab treatment for patients previously treated with bevacizumab
  Interventions: Biological: Dendritic cell vaccination, with optional bevacizumab treatment for patients previously treated with bevacizumab

INTERVENTIONS:
Biological: Dendritic cell vaccination, in addition to standard temozolomide chemotherapy and involved field radiation therapy — Patients will receive a series of four vaccines given weekly during the Induction phase, followed by vaccinations every 8 weeks during the Maintenance phase for as long as patients remain on the study or until the vaccine supply is depleted. In addition to the investigative treatment, patients with newly diagnosed glioblastoma will receive standard temozolomide chemotherapy and radiation treatment, with the vaccine Induction phase beginning at the conclusion of radiation.
  Arms: Cohort A: Patients with newly diagnosed glioblastoma
Biological: Dendritic cell vaccination, with optional bevacizumab treatment for patients previously treated with bevacizumab — Patients will receive a series of four vaccines given weekly during the Induction phase, followed by vaccinations every 8 weeks during the Maintenance phase for as long as patients remain on the study or until the vaccine supply is depleted. Patients with recurrent glioblastoma will not receive additional treatment other than the investigative treatment as long as they remain on study, unless they were previously treated with bevacizumab, in which case they will be allowed to continue receiving bevacizumab
  Arms: Cohort B: Patients with recurrent glioblastoma

SUMMARY:
The purpose of this study is to test the safety and effects of a special type of a cancer vaccine called a 'dendritic cell vaccine' in patients with either newly diagnosed or recurrent glioblastoma. The goal of this dendritic cell vaccine is to activate a patient's own immune system against their tumor. This study utilizes a patient's own immune-stimulating dendritic cells that are isolated in a procedure called leukapheresis. In a laboratory, these dendritic cells are treated in a way that is designed to promote an immune response against cancer stem cells. Then the dendritic cells are injected under the skin in a series of vaccinations, with the goal of activating an immune response against cancer stem cells in the tumor.

To qualify for this study, patients must have very little to no residual tumor visible on a recent MRI. In addition to the vaccines, patients with newly diagnosed glioblastoma will receive standard temozolomide chemotherapy and radiation therapy. Patients with recurrent glioblastoma will not receive any treatment other than the vaccines as long as they are participating in this study, unless they were previously treated with bevacizumab, in which case they will be allowed to continue receiving bevacizumab.

DETAILED DESCRIPTION:
This phase I study for patients with either newly diagnosed or recurrent glioblastoma with minimal residual tumor utilizes a dendritic cell vaccine consisting of autologous dendritic cells that have been pulsed with a lysate derived from an allogeneic glioblastoma stem-like cell line cultured under neurosphere-forming conditions.

Patients will receive a series of four vaccines given weekly during the Induction phase, followed by vaccinations every 8 weeks during the Maintenance phase for as long as patients remain on the study or until the vaccine supply is depleted. In addition to the investigative treatment, patients with newly diagnosed glioblastoma will receive standard temozolomide chemotherapy and radiation treatment, with the Induction phase beginning at the conclusion of radiation. Patients with recurrent glioblastoma will not receive treatment other than the investigative treatment, unless they were previously treated with bevacizumab, in which case they will be allowed to continue receiving bevacizumab.

ELIGIBILITY:
Inclusion Criteria:

1. Cohort A: Newly diagnosed glioblastoma Patients with an initial biopsy or partial resection can qualify for Cohort A if the second surgery (to achieve gross total resection) occurs within 30 days of the initial surgery, without any interval treatment using radiation or chemotherapy between the two surgeries.

   Cohort B: Glioblastoma up to and including third recurrence To qualify for Cohort B, patients must have previously been treated with involved-field radiation therapy with concurrent temozolomide chemotherapy, and pathology from the resection that qualifies the patient for the trial must be consistent with recurrent disease (ie, patients with predominantly pseudoprogression or radiation necrosis are not eligible). Patients who were initially diagnosed with low-grade glioma (ie, WHO grade 2 glioma) with subsequent progression to high-grade glioma are eligible for Cohort B provided they meet all other eligibility criteria. Patients with recurrent high-grade glioma are eligible up to and including third recurrence, and therefore are permitted to have been treated with up to three distinct chemotherapy regimens prior to trial enrollment. Prior and/or continued bevacizumab therapy is allowed.
2. Complete resection of tumor: gross total resection consisting of no gadolinium enhancement or linear gadolinium enhancement along the resection cavity; or subtotal resection consisting of linear enhancement with nodular gadolinium enhancement of less than 1cm x 1cm x 1cm total volume. The qualifying surgical resection must have been performed at Cedars-Sinai in order to allow for tumor stem cell antigen testing.
3. ≥ 18 years of age
4. Karnofsky Performance Score (KPS) of ≥ 70%
5. Baseline hematologic studies and chemistry profiles must meet the following criteria: hemoglobin (Hgb) > 9.9 g/dL, absolute neutrophil count (ANC) > 1000/mm3, platelet count > 100,000/mm3, blood urea nitrogen (BUN) < 30 mg/dL, creatinine < 1.4 mg/dL, alkaline phosphatase (ALP), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 4x upper limit of normal (ULN), prothrombin time (PT) and activated partial thromboplastin time (PTT) ≤ 1.6 x control unless therapeutically warranted
6. Female patients of child bearing potential must have negative serum pregnancy test
7. If not surgically sterile, male and female patients of childbearing age must use double barrier contraception (hormonal; intrauterine device; barrier)
8. Written informed consent, Release of Medical Records Form and HIPAA reviewed and signed by patient or legally authorized representatives
9. Ability to understand and the willingness to sign a written informed consent document.
10. Any Grade 3 or 4 toxicities (according to NCI CTCAE) resolved for at least 2 weeks to Grade 1 or less

Exclusion Criteria:

1. Presence of any other active malignancy or prior history of malignancy that, in the opinion of the Investigator, would interfere with the evaluation of vaccine or interpretation of patient safety or study results.
2. Clinically significant pulmonary, cardiac or other systemic disease that, in the opinion of the Investigator, would interfere with the evaluation of vaccine or interpretation of patient safety or study results - for example:

   1. New York Heart Association > Grade 2 congestive heart failure within 6 months prior to study entry;
   2. Uncontrolled or significant cardiovascular disease, including:

      * Myocardial infarction within 6 months prior to enrollment
      * Uncontrolled angina within 6 months
      * Diagnosed or suspected congenital long QT syndrome
      * Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de pointes);
      * Clinically significant abnormality on electrocardiogram (ECG)
3. Pulmonary disease including or greater than grade 2 dyspnea, laryngeal edema, grade 3 pulmonary edema, pulmonary hypertension according to CTCAE 4.03
4. Severe acute or chronic medical or psychiatric condition that could increase the risk associated with trial participation or trial drug administration or could interfere with the interpretation of trial results and, in the judgment of the investigator, would make the patient inappropriate for entry into the trial. This includes but is not limited to the following: (a) Immunosuppressive disease, (b) Chronic renal disease / failure, (c) Concurrent neurodegenerative disease, (d) Dementia or significantly altered mental status that would prohibit the understanding or rendering of informed consent and compliance with the requirements of the protocol.
5. Presence of an acute infection requiring active treatment with antibiotics/antivirals; prophylactic administration is allowed
6. Active autoimmune disorder or known history of an autoimmune neurologic condition (e.g. Guillain-Barre syndrome). Patients with vitiligo, type 1 diabetes mellitus, hypothyroidism due to autoimmune condition only requiring hormone replacement therapy, psoriasis not requiring systemic therapy, or conditions not expected to recur in the absence of an external trigger are permitted to enroll.
7. Known human immunodeficiency virus positivity or acquired immunodeficiency syndrome related illness or other serious medical condition
8. Breastfeeding
9. Received any other therapeutic investigational agent within 30 days of enrollment
10. Contraindication to MRI
11. Foreseeable condition which would preclude the reduction of steroids (dexamethasone) to a maximum of 2 mg BID within a week prior to apheresis.
12. Any foreseeable scheduling constraint that would prevent a patient in Cohort A from starting chemoradiation within 7 weeks of surgery, and any foreseeable scheduling constraint that would prevent a patient in Cohort B from starting the Vaccine Induction Phase within 7 weeks of surgery.
13. Any concomitant chemotherapy other than standard-dose temozolomide for patients in Cohort A; any concomitant chemotherapy for patients in Cohort B, with the exception of the antiangiogenic humanized monoclonal antibody bevacizumab, which is allowed for patients treated with bevacizumab prior to enrollment in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2014-01-08 (Actual); Primary Completion 2019-01-23 (Actual); Study Completion 2021-07-10 (Actual)

PRIMARY OUTCOMES:
Assess safety and tolerability according to National Cancer Institute Common Toxicity Criteria for Adverse Events (NCI CTCAEs) Version 4.03 | 1 year
Assess the number of serious adverse events | 1 year
Assess treatment-related toxicities | 1 year
  We will assess possible vaccine-related adverse effects, including but not limited to cerebral edema, autoimmune reactions, and allergic reactions.

SECONDARY OUTCOMES:
Evaluate Overall Survival (OS) and Progression-Free Survival (PFS) | 2 years
Evaluate health-related quality of life parameters | 2 years
Assess the overall response rate, defined as the percentage of patients showing either partial response or complete response, in patients with subtotal resection | 2 years
Evaluate immune response by assessing cytotoxic T cell activity in vitro pre- vs post-vaccination | 2 years
Assess tumor stem cell antigen expression | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jethro Hu, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

REFERENCES:
- [Derived] Hu JL, Omofoye OA, Rudnick JD, Kim S, Tighiouart M, Phuphanich S, Wang H, Mazer M, Ganaway T, Chu RM, Patil CG, Black KL, Shiao SL, Wang R, Yu JS. A Phase I Study of Autologous Dendritic Cell Vaccine Pulsed with Allogeneic Stem-like Cell Line Lysate in Patients with Newly Diagnosed or Recurrent Glioblastoma. Clin Cancer Res. 2022 Feb 15;28(4):689-696. doi: 10.1158/1078-0432.CCR-21-2867. PMID 34862245